CLINICAL TRIAL: NCT01387191
Title: Drug Use Investigation for FLOLAN (Epoprostenol) Injection 0.5mg・1.5mg
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 112300
Record Dates: First submitted 2011-06-30; First posted 2011-07-04 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Epoprostenol

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subjects prescribed epoprostenol: Subjects with pulmonary arterial hypertension prescribed epoprostenol injection during study period
  Interventions: Drug: Epoprostenol

INTERVENTIONS:
Drug: Epoprostenol

SUMMARY:
The objective of this study is to evaluate the incidence of adverse events in Japanese pulmonary arterial hypertension subjects treated with epoprostenol injection based on prescribing information under the conditions of general clinical practice and also to grasp the following items;

1. Unknown adverse reactions (especially, significant adverse reactions)
2. Adverse reaction onset status under practical drug use conditions
3. Factors possibly influential on safety
4. Factors possibly influential on efficacy
5. Patient's prognosis, efficacy and safety in long-term use

ELIGIBILITY:
Inclusion Criteria:

* Subjects with cardiovascular disease

Exclusion Criteria:

* Subjects with hypersensitivity to epoprostenol
* Subjects with right cardiac failure during an acute exacerbation
* Subjects with severe left ventricular systolic dysfunction
* Subjects with serious left ventricular dysfunction
* Subjects whose pulmonary edema getting worse during dose initiation

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All Japanese subjects with pulmonary arterial hypertension who are treated with epoprostenol injection
Sampling Method: Probability Sample
Enrollment: 748 (Actual)
Dates: Start 1999-08; Primary Completion 2009-04 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
The number of incidence of adverse events in Japanese subjects with pulmonary arterial hypertension treated with epoprostenol injection | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline